CLINICAL TRIAL: NCT05944016
Title: DOUBLE PRO-TECT Alport: a Confirmatory, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Effect of Dapagliflozin on the Progression of Chronic Kidney Disease in Adolescents and Young Adult Patients with Alport Syndrome
Brief Title: Phase 3 Clinical Trial with Dapagliflozin in Chronic Kidney Disease in Adolescents and Young Adult Patients
Acronym: DOUBLE_PROTECT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Goettingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Prof. Dr. O. Gross, Prof. Dr. Oliver Gross, University Hospital Goettingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMG DOUBLE PRO-TECT 2023
Record Dates: First submitted 2023-07-01; First posted 2023-07-13 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Failure in Children and Young Adults
Keywords: chronic kidney disease in children; pediatric population; nephroprotective therapy in children; Alport syndrome; type IV collagen disease
MeSH Terms: conditions — Nephritis, Hereditary | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Experimental intervention: Dapagliflozin (standard dose 10 mg p.o. once daily). Control intervention: Placebo therapy.
Who Masked: Participant, Investigator
Masking Description: double-blinded study using capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin (standard dose 10 mg p.o. once daily).
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin (standard dose 10 mg p.o. once daily)
  Arms: Dapagliflozin
Drug: Placebo — Placebo (standard dose p.o. once daily)
  Arms: Placebo

SUMMARY:
Recent trials have demonstrated positive renal outcomes of sodium-glucose co-transporter-2 inhibitors (SGLT2i) additive to angiotensin-converting-enzyme inhibitors (ACEis) in adult patients with diabetic and non-diabetic chronic kidney disease (CKD). These trials included no children. The hypothesis of DOUBLE PRO-TECT Alport is to demonstrate superiority of the SGLT2i dapagliflozin in preventing progression of the chronic kidney disease Alport syndrome in children and young adults at early stages of disease. Preventing the rise of albuminuria by dapagliflozin would result in a very significant delay of end-stage kidney failure (ESKF) and improved quality of life. If successful, DOUBLE PRO-TECT Alport will change the treatment recommendations for children with CKD, who have a very high unmet medical need.

ELIGIBILITY:
Key inclusion criteria:

Early stages of CKD with established diagnosis of Alport syndrome at visit 1 (screening)

* adolescents ≥ 10 to < 18 years with albuminuria (UACR ≥ 300mg/g creatinine) AND
* eGFR ≥ 30 ml/min/1.73 m2 OR
* adults ≥ 18 to < 40 years with albuminuria (UACR ≥ 500mg/g creatinine) AND
* eGFR ≥ 60 ml/min/1.73 m2

  1. Molecular-genetic diagnosis or diagnosis established by kidney biopsy
  2. Stable RAS blockade as background therapy.
  3. Signed and dated written informed consent.

Key exclusion criteria:

1. Medical history that might limit the individual's ability to take trial treatments.
2. Treatment with any SGLT2 inhibitor or within 4 weeks prior to Visit 1.
3. eGFR<60 mL/min/1.73 m2 (CKD-EPI) or requiring dialysis or after kidney-transplantation
4. Uncontrolled arterial hypertension (blood pressure above 145/95 mmHg).
5. Known hypersensitivity or allergy to the investigational products.
6. Any previous or current alcohol or drug abuse.
7. Participation in another trial with an investigational drug ongoing.
8. Women, who are nursing or pregnant, or who are not practicing an acceptable method of birth control.

Ages: 10 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 48 weeks
  Change from baseline urine albumin to creatinine ratio (UACR) after 48 weeks

SECONDARY OUTCOMES:
Key secondary efficacy endpoint | 52 weeks
  Change from baseline estimated glomerular filtration rate (eGFR) after 52 weeks (4 weeks off treatment)
Key secondary safety endpoint | 52 weeks
  Adverse events (including serious adverse events)
Adverse events (AE) of special interest | 52 weeks
  (a) Ketoacidosis or symptomatic hypoglycemic event.
Adverse events (AE) of special interest | 52 weeks
  (b) Hyperkalemia (potassium levels ≥15% of the upper normal limit)
Adverse events (AE) of special interest | 52 weeks
  (c) Decline in eGFR of ≥ 30% relative from baseline eGFR.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gross, MD, Principal Investigator — University Medicine Goettingen, Germany
Locations (16):
- Germany (16):
  - Universitätsklinikum Heidelberg - Children, Heidelberg, Baden-Württenberg
  - LMU Klinikum, München, Bavaria
  - v. Haunersches Kinderhospital, München, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf - Adults, Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf - Children, Hamburg, Hamburg
  - Clementine Kinderhospital, Frankfurt am Main, Hesse
  - University Medicine Goettingen - Adults, Göttingen, Lower Saxony
  - University Medicine Goettingen - Childrens Hospital, Göttingen, Lower Saxony
  - Universitätsklinik Köln - Adults, Cologne, North Rhine-Westphalia
  - Universitätsklinik Köln - Children, Cologne, North Rhine-Westphalia
  - Universitätsklinik Münster - Adults, Münster, North Rhine-Westphalia
  - Universitätsklinikum Münster - Children, Münster, North Rhine-Westphalia
  - Universitätsklinik Leipzig - Children, Leipzig, Saxony
  - Universitätsklinikum Leipzig - Adults, Leipzig, Saxony
  - Charite Berlin - Adults, Berlin, State of Berlin
  - Charite Berlin - Children, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after end of study on request and with valid IRB-vote and data protection protocol by applicant.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Documents will be shared after end of study on request and with valid IRB-vote and data protection protocol by applicant.
Access Criteria: IPD will be shared after end of study on request and with valid IRB-vote and data protection protocol by applicant.

REFERENCES:
- [Background] Gross O, Boeckhaus J, Weber LT, Heerspink HJL, Simon JF, Ahmed R, Gerst C, Duerr U, Walker F, Tostmann R, Helm J, Asendorf T, Friede T; study group of the German Society of Pediatric Nephrology. Protocol and rationale for a randomized controlled SGLT2 inhibitor trial in paediatric and young adult populations with chronic kidney disease: DOUBLE PRO-TECT Alport. Nephrol Dial Transplant. 2025 Apr 1;40(4):679-687. doi: 10.1093/ndt/gfae180. PMID 39122650
- [Background] Gross O, Haffner D, Schaefer F, Weber LT. SGLT2 inhibitors: approved for adults and cats but not for children with CKD. Nephrol Dial Transplant. 2024 May 31;39(6):907-909. doi: 10.1093/ndt/gfae029. No abstract available. PMID 38308509